CLINICAL TRIAL: NCT00030264
Title: Vinblastine/Methotrexate For Severe Progressive Plexiform Neurofibromas: A Phase II Study
Brief Title: Combination Chemotherapy in Treating Patients With Neurofibromatosis and Progressive Plexiform Neurofibromas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-2339; CHP-686 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Neurofibromatosis Type 1; Precancerous Condition
Keywords: plexiform neurofibroma; neurofibromatosis type 1
MeSH Terms: conditions — Neurofibromatosis 1; Precancerous Conditions; Neurofibroma, Plexiform | interventions — Methotrexate; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methotrexate & Vinblastine (Experimental): Methotrexate and Vinblastine will be given once a week for the first 26 weeks and then every two weeks for the next 26 weeks or until disease progression (whichever occurs first).
  Interventions: Drug: Methotrexate; Drug: Vinblastine

INTERVENTIONS:
Drug: Methotrexate — Methotrexate will be given at a dose of 30mg/m2/week intramuscular (IM) or intravenous (IV) for the first 26 weeks, then every 2 weeks for the next 26 weeks or until disease progression (whichever occurs first)
Drug: Vinblastine — Vinblastine will be given at a dose of 6mg/m2/week intravenous (IV) for for the first 26 weeks, then every 2 weeks for the next 26 weeks or until disease progression (whichever occurs first). Maximum actual dose may not exceed 10mg.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining methotrexate with vinblastine may be effective treatment for neurofibromatosis type 1 associated with progressive plexiform neurofibromas.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have neurofibromatosis type 1 associated with progressive plexiform neurofibromas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of chronic vinblastine and methotrexate on time to disease progression in children or young adults with progressive plexiform neurofibroma associated with neurofibromatosis type 1.
* Determine the objective response rate in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: Patients are stratified according to tumor status (severely debilitating and/or life-threatening vs cosmetically disfiguring).

Patients receive methotrexate and vinblastine IV weekly for 26 weeks and then every 2 weeks for 26 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 3 months during study participation.

Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study within approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Progressive, debilitating, severely disfiguring or life-threatening plexiform neurofibroma (PN) which is not surgically resectable and for which there is no other standard medical management. Histologic confirmation of tumor is not required in the presence of consistent clinical and radiographic findings. However, if any clinical observation or scan suggests possible malignant transformation, the tumor must be biopsied prior to therapy. In addition to PN, all study subjects must have at least one other diagnostic criteria for Neurofibromatosis type 1 (NF1) listed below:

   * 6 or more café-au-lait spots > 0.5 cm in prepubertal subjects or > 1.5 cm in postpubertal subjects
   * freckling in the axilla or groin
   * optic glioma
   * 2 or more lisch nodules
   * a distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
   * a first degree relative with NF1
2. Adequate bone marrow, renal, hepatic function:

   * Absolute Neutrophil Count (ANC)> 1000 and platelet count >100,000 prior to initiation of therapy
   * must have normal renal function: Blood Urea Nitrogen (BUN)/Creatinine <1.5x normal for age), alkaline phosphatase (ALP), albumin, total protein and bilirubin
   * must have normal liver function: Bilirubin, alanine transaminase (ALT), aspartate aminotransferase (AST) < 1.5x normal for age
3. Patients must have measurable PN by direct physical examination (documented by clinical measurement of tumor and serial photography) or by imaging studies. Most patients will have tumors that can be measured by magnetic resonance imaging (MRI), however, some patients may have cosmetically disfiguring PN which would be best measured clinically and with serial photography throughout treatment and follow-up. A measurable lesion is one whose size can be quantified in at least 2 dimensions. There must be evidence of recurrent or progressive disease as documented by an increase in size or the presence of new lesions on MRI. Progression is defined as the appearance of new tumors or a measurable increase in the sum of the product of the two longest perpendicular diameters of the index lesion(s) over a time period < 12 months prior to evaluation for this study. For purposes of this study, index PN lesions will be those PNs evaluated as the most life-threatening, debilitating, cosmetically disfiguring, and/or most easily measured.
4. Prior therapy: Patients with NF1 are eligible at the time of recurrence or progression of inoperable PN. A surgical consultation should be obtained prior to enrollment on the study to evaluate if tumor resection is a feasible option. Patients will only be eligible if complete tumor resection is not feasible or if a patient with a surgical option refuses surgery. Since there is no standard effective chemotherapy for patients with NF1 and progressive PN, patients may be treated on this trial without having received prior therapy. Patients must have recovered from the toxic effects of all prior therapy before entering this study. The Cancer Therapy Evaluation Program Common Toxicity Criteria (CTC) Version 2.0 will be used for toxicity assessment. Recovery is defined as a toxicity grade < 2, unless otherwise specified in the Inclusion and Exclusion Criteria. Patients must have had their last dose of radiation therapy at least 6 weeks prior to study entry, and their last dose of chemotherapy at least four weeks prior to study entry. Patients who received granulocyte-colony stimulating factor (G-CSF) after the prior cycle of chemotherapy must be off G-CSF for at least one week prior to entering this study.
5. Performance status: Patients should have a life expectancy of at least 12 months and a Lansky or Karnofsky performance score of > 60. Patients who are wheelchair bound because of paralysis should be considered "ambulatory" when they are mobile and active in their wheelchairs rather than actually ambulatory.
6. A Pregnancy test must be negative for females of childbearing age.
7. Informed consent: All patients or their legal guardians (if the patient is less than 18 years old) must sign an approved document of informed consent indicating their understanding of the investigational nature and the risks of this study before beginning therapy. When appropriate pediatric patients will be included in all discussion in order to obtain verbal assent.

Exclusion Criteria:

1. Pregnant females are excluded
2. Patient has had treatment with an investigational agent within the past 30 days.
3. Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the tumor or immunotherapy.
4. Inability to return for follow-up visits or obtain follow-up studies required to assess toxicity and response to therapy.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2001-02; Primary Completion 2013-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean B. Belasco, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 eligible subjects were enrolled at the Children's Hospital of Philadelphia and Texas Children's Hospital between March 2001 and June 2011
Period: Overall Study
Arm/Group | Methotrexate & Vinblastine
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Methotrexate & Vinblastine
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 5.56 [0.34 to 23.99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: Disease progression was assessed both radiographically and clinically.
  Tumor assessments to assess for radiographic disease progression were assessed by magnetic resonance imaging (MRI) measurement whenever possible or computed tomography (CT) scan and/or tumor measurement during physical examination of palpable lesions. Clinical assessments for clinical progression of disease were assessed by treating physician or designee.
  Progressive disease as measured by the appearance of new lesions; an increased size of index tumor(s) by >/= 25% of the sum of the products of baseline measurements; and/or by increase in symptoms.
Time Frame: 6 months
Population: 20 subjects were analyzed for time to progression. 3 subjects were not included in the response analysis due to lost to follow up (N=2) or progression of comorbid condition which required early termination (N=1)
Measure: Mean (Full Range); unit: Months
Arm/Group | Methotrexate & Vinblastine
Number analyzed (Participants) | 20
Months
  Total | 25.8 [0.2 to 85.0]
  Radiographic Progression: number analyzed (Participants) | 6
  Radiographic Progression | 29.2 [3.1 to 58.5]
  Clinical Progression: number analyzed (Participants) | 14
  Clinical Progression | 25.8 [0.2 to 85.0]

ADVERSE EVENTS:
Description: For non-serious events, CTCAE Grade 3 and 4 were collected.
Arm/Group | Methotrexate & Vinblastine
All-Cause Mortality (participants affected / at risk) | 3/23
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate & Vinblastine (N=23)
Infection - Bacterial (Infections and infestations) | 1 (1) — Fever, otitis externa, otitis media, cellulitis
Hepatic - Other - Cholecytitis (Hepatobiliary disorders) | 1 (1) — Acute cholecystitis with fever, nausea and vomiting, elevated liver tests
Anorexia (Gastrointestinal disorders) | 1 (1)
Pulmonary - Other - Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection - Viral (Infections and infestations) | 1 (1) — Parainfluenza with grade 4 ANC
Febrile neutropenia (Investigations) | 1 (1) — fever with neutropenia
Fever (Investigations) | 1 (1) — Fever with upper respiratory infection symptoms
Fever (Investigations) | 1 (1) — Fever NOS
Infection (Infections and infestations) | 1 (1) — Chicken Pox
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate & Vinblastine (N=23)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8 (15)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Infection - Viral (Infections and infestations) | 1 (1) — Parainfluenza
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 1 (1) — ALT increased

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes